CLINICAL TRIAL: NCT04804943
Title: Pilot Clinical Study to Investigate the Efficacy and Safety of NOA-001 for the Treatment of Patients With Acute Respiratory Distress Syndrome.
Brief Title: Pilot Clinical Study of NOA-001 for ARDS (Acute Respiratory Distress Syndrome)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOA001ARDS01
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: COVID-19; Diffuse Alveolar Damage; DAD; Acute Respiratory Distress Syndrome; ARDS; NOA-001; Hemoperfusion
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NOA-001 group (ARDS caused by Non-COVID-19 cohort) (Experimental): Patients will receive the standard and NOA-001 therapy.
  Interventions: Device: NOA-001
- Standard treatment group (ARDS caused by Non-COVID-19 cohort) (No Intervention): Patients will receive the standard therapy.
- NOA-001 group (ARDS caused by COVID-19 cohort) (Experimental): Patients will receive the standard and NOA-001 therapy.
  Interventions: Device: NOA-001

INTERVENTIONS:
Device: NOA-001 — NOA-001 will be replaced regularly (at 22 to 24 hours after the initiation of procedure), and will be continuously performed until 168 hours from the enrollment.
  Arms: NOA-001 group (ARDS caused by COVID-19 cohort); NOA-001 group (ARDS caused by Non-COVID-19 cohort)

SUMMARY:
The primary object of this clinical study is to investigate the efficacy and the safety of NOA-001 in patients with ARDS (ARDS caused by Non-COVID-19 or COVID-19).

DETAILED DESCRIPTION:
(ARDS caused by Non-COVID-19 cohort): The objectives of this clinical study is to investigate the efficacy and safety of NOA-001 in patients with ARDS caused by Non-COVID-19. The number of patients enrolled is 30 (20 patients in the NOA-001 group and 10 patients in the standard therapy group).

(ARDS caused by COVID-19 cohort): The objectives of this clinical study is to investigate the efficacy and the safety of NOA-001 in patients with ARDS caused by COVID-19. The number of patients enrolled is 15 (in the NOA-001 group only).

ELIGIBILITY:
(ARDS caused by Non-COVID-19 cohort)

Inclusion Criteria:

At Informed Consent

1. Patients with ARDS confirmed by the Berlin definition based on the following diagnostic criteria (a)-(d):

   1. Patients within 7 days from invasion or exacerbation of respiratory symptoms or acute onset of ARDS.
   2. Patients with respiratory failure not fully explained by cardiac failure or fluid overload; Need objective assessment (e. g., echo-cardiography) to exclude hydrostatic edema if no risk factor present
   3. Patients with bilateral opacities not fully explained by effusions, lobar/ lung collapse, or nodules on chest X-ray or CT scan
   4. Patients with PaO2/ FiO2 ratio ≤ 300 mmHg (PEEP ≥ 5 cmH2O)
2. Patients who are intubated and mechanically ventilated
3. Patients who can be enrolled in the study within 96 hours after initiation of mechanical ventilation
4. Patients aged ≥ 16 years at informed consent (Signed informed consent form from legally acceptable representative must be available if patient is aged < 20 years)

At Enrollment

1. Patients with PaO2/ FiO2 ratio ≥ 50 mmHg and ≤ 200 mmHg (PEEP ≥ 5 cmH2O)
2. Patients with bilateral opacities not fully explained by effusions, lobar/ lung collapse, or nodules on CT scan within 48 hours before enrollment
3. Patients who are intubated and mechanically ventilated
4. Patients who can be enrolled in the study within 96 hours after initiation of mechanical ventilation

Exclusion Criteria:

At Informed Consent

1. Patients who are considered to be extremely unlikely to withdraw from mechanical ventilation
2. Patients who are treated with ECMO or HFOV
3. Patients with renal dialysis therapy for chronic renal failure
4. Patients with congestive heart failure (NYHA class IV)
5. Patients with acuter left ventricular failure
6. Patients with liver failure (Child-Pugh grade C)
7. Patients who have burns in excess of 15% total body surface area
8. Patients after resuscitation from cardiac arrest
9. Patients with a history of hypersensitivity to the anticoagulants (Heparin or Nafamostat mesylate)
10. Patients who have received cytapheresis, blood purification therapy with cytokine adsorbing devices or endotoxin removal therapy within 7 days prior to informed consent
11. Patients with pregnancy or lactating
12. Patients tested positive for COVID-19

At Enrollment

1. Patients who are considered to be extremely unlikely to withdraw from mechanical ventilation
2. Patients who are treated with ECMO or HFOV after obtaining informed consent prior to enrollment
3. Patients with platelet count ≤ 50,000 /mm3 by the latest blood test
4. Patients who have received cytapheresis, blood purification therapy with cytokine adsorbing devices or endotoxin removal therapy between informed consent and enrollment
5. Patients whose life expectancy is ≤ 24 hours after enrollment
6. Patients after resuscitation from cardiac arrest between informed consent and enrollment
7. Patients tested positive for COVID-19 between informed consent and enrollment

(ARDS caused by COVID-19 cohort)

Inclusion Criteria:

At Informed Consent

1. Patients tested positive for COVID-19
2. Patients with ARDS confirmed by the Berlin definition based on the following diagnostic criteria (a)-(d):

   1. Patients within 7 days from invasion or exacerbation of respiratory symptoms or acute onset of ARDS.
   2. Patients with respiratory failure not fully explained by cardiac failure or fluid overload; Need objective assessment (e. g., echo-cardiography) to exclude hydrostatic edema if no risk factor present
   3. Patients with bilateral opacities not fully explained by effusions, lobar/ lung collapse, or nodules on chest X-ray or CT scan
   4. Patients with PaO2/ FiO2 ratio ≤ 300 mmHg (PEEP ≥ 5 cmH2O)
3. Patients who are intubated and mechanically ventilated
4. Patients who can be enrolled in the study within 96 hours after initiation of mechanical ventilation
5. Patients aged ≥ 16 years at informed consent (Signed informed consent form from legally acceptable representative must be available if patient is aged < 20 years)

At Enrollment

1. Patients with PaO2/ FiO2 ratio ≥ 50 mmHg and ≤ 200 mmHg (PEEP ≥ 5 cmH2O)
2. Patients who are intubated and mechanically ventilated
3. Patients who can be enrolled in the study within 96 hours after initiation of mechanical ventilation

Exclusion Criteria:

At Informed Consent

1. Patients who are considered to be extremely unlikely to withdraw from mechanical ventilation
2. Patients who are treated with ECMO or HFOV
3. Patients with renal dialysis therapy for chronic renal failure
4. Patients with congestive heart failure (NYHA class IV)
5. Patients with acuter left ventricular failure
6. Patients with liver failure (Child-Pugh grade C)
7. Patients who have burns in excess of 15% total body surface area
8. Patients after resuscitation from cardiac arrest
9. Patients with a history of hypersensitivity to the anticoagulants (Heparin or Nafamostat mesylate)
10. Patients who have received cytapheresis, blood purification therapy with cytokine adsorbing devices or endotoxin removal therapy within 7 days prior to informed consent
11. Patients with pregnancy or lactating

At Enrollment

1. Patients who are considered to be extremely unlikely to withdraw from mechanical ventilation
2. Patients who are treated with ECMO or HFOV after obtaining informed consent prior to enrollment
3. Patients with platelet count ≤ 50,000 /mm3 by the latest blood test
4. Patients who have received cytapheresis, blood purification therapy with cytokine adsorbing devices or endotoxin removal therapy between informed consent and enrollment
5. Patients whose life expectancy is ≤ 24 hours after enrollment
6. Patients after resuscitation from cardiac arrest between informed consent and enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
Ventilator Free Days (VFD, Days alive and ventilator-free) | Day 28
  VFD is a composite measure of all-cause mortality and the number of days free of mechanical ventilation (VFD) within 28 days.

SECONDARY OUTCOMES:
All-cause Mortality | Up to Day 28, 60 and 90
  Fatalities, mortality all-causes
Mortality in ICU | Up to Day 28
  All-cause mortality for patients who died in Intensive Care Units.
Mortality in Hospital | Up to Day 28
  The number of patients who died in hospital
Changes in PaO2/ FiO2 ratio | Up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Showa University Hospital, Tokyo, Japan